CLINICAL TRIAL: NCT00509301
Title: Open-label Dose Confirmation and Dosimetry Study of Interstitial 131I-chTNT-1/B MAb (Cotara®) for the Treatment of Recurrent Glioblastoma Multiforme
Brief Title: Safety & Radiation Distribution Study of Cotara® in Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Jennifer Lai, MBA, CCRA, Peregrine Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0602; NCT00516789 (obsolete NCT alias)
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: brain cancer; Cotara; radioactive isotope; monoclonal antibody; radiation distribution
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — 131I-chimeric TNT-1-B monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 1.5 mCi/cc
  Interventions: Drug: 131-I-chTNT-1/B MAB
- 2 (Experimental): 2.0 mCi/cc
  Interventions: Drug: 131-I-chTNT-1/B MAB
- 3 (Experimental): 2.5 mCi/cc
  Interventions: Drug: 131-I-chTNT-1/B MAB

INTERVENTIONS:
Drug: 131-I-chTNT-1/B MAB — The study drug is given interstitially for approximately 25 hours at a dose of 1.5, 2.0, or 2.5 mCi/cc.
  Other Names: Cotara

SUMMARY:
RATIONALE: Cotara® is an experimental new treatment that links a radioactive isotope (iodine 131) to a targeted monoclonal antibody. This monoclonal antibody is designed to bind tumor cells and deliver radiation directly to the center of the tumor mass while minimizing effects on normal tissues. Cotara® thus literally destroys the tumor "from the inside out." This may be an effective treatment for glioblastoma multiforme, a malignant type of brain cancer.

PURPOSE: This trial is studying the safety and radiation distribution of Cotara® in patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To confirm the dose limiting toxicities (DLT) and maximum tolerated dose (MTD) of 131I-chTNT-1/B MAb (Cotara®) when given as a single 25 hour interstitial infusion in patients with recurrent GBM
* To characterize the biodistribution and radiation dosimetry of Cotara®

OUTLINE:

This is an open-label, dose escalation study of Cotara®.

All patients will receive 3 mCi of Cotara® for biodistribution and radiation dosimetry purposes. In addition, patients will receive escalating therapeutic dose levels of Cotara® for confirmation of the maximum tolerated dose (MTD). After completion of study treatment, patients are followed for a minimum of 12 weeks and until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent GBM
* Patients with a Clinical Target Volume between 5 and 60 cc (inclusive)
* Patients of 18 years of age or older
* Karnofsky Performance Status ≥ 60 at screening
* Patients not on steroids or maintained on a stable corticosteroid regimen (± 4 mg) for at least 2 weeks prior to study entry

Exclusion Criteria:

* Patients with infratentorial tumor(s), exophytic intra-ventricular tumor(s) or subependymal tumor spread extending greater than 2 cm
* Patients with diffuse disease
* Patients with known or suspected allergy to study medication or iodine
* Patients who received investigational agents within 30 days prior to baseline
* Patients who received surgical resection within 4 weeks from baseline
* Patients with known HIV or evidence of active hepatitis
* Patients who cannot undergo MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To confirm dose limit and maximum tolerated dose and to characterize radiation distribution

CONTACTS AND LOCATIONS:
Overall Officials: Sunil J Patel, MD, Principal Investigator — Medical University of South Carolina; Kenneth M Spicer, MD PhD, Principal Investigator — Medical University of South Carolina; Kevin D Judy, MD, Principal Investigator — University of Pennsylvania; William R Shapiro, MD, Principal Investigator — Barrow Neurological Institute; Andrew E Sloan, MD, FACS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (4):
- United States (4):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina